CLINICAL TRIAL: NCT03512574
Title: The Effect of the Combination of Pregabalin and Dexmedetomidine on the Management of Postoperative Pain in Patients Undergoing Total Knee Arthroplasty (TKA) or Total Hip Arthroplasty (THA) Under Spinal Anesthesia
Brief Title: Combination Effects of Pregabalin and Dexmedetomidine on Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee, Professor,M.D.,Ph.D, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WonkwangUH5
Record Dates: First submitted 2018-04-08; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative
Keywords: pregabalin, dexmedetomidine, postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group PD (Experimental): combination of pregabalin and dexmedetomidine
  Interventions: Drug: Pregabalin and dexmedetomidine
- Group P (Active Comparator): pregabalin +placebo
  Interventions: Drug: Pregabalin
- Group D (Active Comparator): placebo + dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Group C (Placebo Comparator): placebo + placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pregabalin — One hour before spinal anesthesia, patients received pregabalin 150 mg capsule orally and the same calculated volume of normal saline till completion of the surgery
  Other Names: Lyrica
  Arms: Group P
Drug: Dexmedetomidine — One hour before spinal anesthesia, patients received placebo and a bolus dose of 0.5 μg /kg IV dexmedetomidine was given over 10 min before induction of spinal anesthesia, a bolus dose of 0.5 μg /kg IV till completion of the surgery
  Other Names: precedex
  Arms: Group D
Other: Placebo — One hour before spinal anesthesia, patients received placebo and the same calculated volume of normal saline till completion of the surgery
  Arms: Group C
Drug: Pregabalin and dexmedetomidine — One hour before spinal anesthesia, patients received pregabalin 150 mg orally and a bolus dose of 0.5 μg /kg IV dexmedetomidine was given over 10 min before induction of spinal anesthesia, a bolus dose of 0.5 μg /kg IV till completion of the surgery.
  Other Names: study drugs
  Arms: Group PD

SUMMARY:
Pregabalin and dexmedetomidine have been introduced to manage postoperative pain. The present study aimed to evaluate the effect of the combination of two drugs on pain relief in patients undergoing total knee or hip arthroplasty under spinal anesthesia

DETAILED DESCRIPTION:
One hundred and twenty-four patients undergoing total knee or hip arthroplasty under spinal anesthesia were randomly assigned to either group C (n = 31, placebo), group P (n = 33, pregabalin), group PD (n = 29, pregabalin and dexmedetomidine) or group D (n = 31, dexmedetomidine). One hour before spinal anesthesia, patients received pregabalin 150 mg or placebo orally and a bolus dose of 0.5 μg /kg IV dexmedetomidine was given over 10 min before induction of spinal anesthesia, followed by a continuous infusion of 0.5 μg/kg/hr or the same calculated volume of normal saline till completion of the surgery. Clinically relevant pain for 24 h after surgery including time to first analgesic request visual analog scale (VAS), ketorolac dose, and patient controlled analgesics (PCA) volume consumed were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Aged 18-75 years

One hundred and twenty-four patients with intact cognitive function to understand this study undergoing elective total knee or hip arthroplasty under spinal anesthesia

Exclusion Criteria:

* Pregnant
* Allergic and/or contraindicated to the study drugs
* American Society of Anesthesiologists (ASA) score III and above
* Having drug
* Alcohol addiction
* Renal failure
* Diabetes mellitus
* Epilepsy
* currently using opioids for chronic pain and/or any of the drugs studied.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Patient controlled analgesics (PCA) volume | For 24 hours
  Patient controlled analgesics (PCA) volume consumed for 24 hours after surgery

SECONDARY OUTCOMES:
time to first analgesic request | for 24 hours
  time to first analgesic request for 24 hours after surgery
visual analog scale (VAS) | for 24 hours
  The VAS consisted of a straight line with the left end of the line representing no pain and the right end of the line representing the worst pain. Patients were asked to mark the position on the line corresponding to their perception of pain. The VAS scores for pain at rest and on movement were measured at intervals of 24, and 48 hours after surgery
ketorolac dose | for 24 hours
  ketorolac dose for 24 hours after surgery
adverse effects | within the first 24 hours postoperatively
  Perioperative adverse effects Shivering, blurred vision, headache, dizziness, dry mouth, nausea/vomiting during the first 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Gilho Lee, M.D., Principal Investigator — Wonkwang University Hospital
Locations (1):
- WonwangUH, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No